CLINICAL TRIAL: NCT04294303
Title: Heart Failure Self-Management Using a Mobile Web-Based Telemonitoring System- Impact on Hospital Readmissions and Quality of Life SELF-e HF
Brief Title: Use of Telemonitoring System in Heart Failure Patients
Acronym: I get better
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danbury Hospital (Other)
Responsible Party: Principal Investigator, Ira Galin, Associate Director of the vascular Medicine Program, Danbury Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-608
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure; Quality of Life
MeSH Terms: conditions — Heart Failure | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Experimental): Subjects were assigned to web based telemonitoring system.
  Interventions: Other: web based telemonitoring system
- Control (Other): Subjects were assigned to conventional monitoring.
  Interventions: Other: Conventional

INTERVENTIONS:
Other: web based telemonitoring system — Subjects in the telemonitoring group were given an iPad with installed iHealth application, a scale, and an electronic blood pressure monitor (a mobile web-based telemonitoring system). These devices were interconnected via Bluetooth. The iPad had permanent internet connection. Patients were taught to use the equipment to check and record their weight, blood pressure, and heart rate every morning, for 45 days after the hospital discharge. Data was automatically uploaded via iHealth application in a secure database.
  Arms: Telemonitoring
Other: Conventional — Subjects in the control group received the standard patient teaching, including an instruction to self-monitor their weight.
  Arms: Control

SUMMARY:
Heart failure is a major public health problem worldwide. Heart failure is one of the most common causes for hospitalizations among people over 65 years of age in the United States. Nationwide, approximately 25% of patients admitted to a hospital for heart failure are readmitted to a hospital within 30 days.Multiple transitional care interventions, including telemonitoring, aimed to decrease hospital readmission rates and improve quality of life in heart failure (HF) patients have been explored. Most studies evaluated effectiveness of telemonitoring used in conjunction with other interventions. In this study, investigators studied the role of a potentially cost-effective, telemonitoring program in reducing readmissions and improving quality of life among patients admitted with HF exacerbation in a teaching hospital. They aimed to determine impact of a standalone telemonitoring system.

Primary outcome: Rate of hospital readmission for heart failure Secondary outcomes: Quality of life, Perceived effect of the intervention on heart-failure related care

DETAILED DESCRIPTION:
60 patients will be recruited for this study. After signing the consent form, participant will be randomized to receive usual care (i.e. they will get the current standard care for patients with heart failure) or usual care and participation in the iGetBetter program. Participant will complete a questionnaire in the hospital about their quality of life. iGetBetter group will be given a Bluetooth-equipped scale, blood pressure cuff, and a tablet with a data plan. Participant will check their weight and blood pressure at home daily, using the equipment provided. This information will be sent via the internet to iGetBetter's web server, where the data will be temporarily stored. The data will be monitored by the physician researcher. If their blood pressure is high (e.g. greater than or equal to 140/90 for two days in a row) or they gain a significant amount of weight (e.g. 2 pounds in two days), the study team will be automatically notified. A member of the study team will alert participant cardiologist and the cardiologist will have the option to make any recommendations, such as contacting the subject to schedule an office visit.

Total participation in this study will last 45 days after patient is discharged from the hospital.

Regardless of the assigned group, participant will be asked to complete two questionnaires after 45 days. A member of the research team will contact participant by phone to complete these questionnaires. One of these questionnaires will investigate their quality of life; the other will assess how participant feel the care they have received has affected their health. Patients assigned to the iGetBetter group will also complete a third survey about their satisfaction with the program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Admitted to Danbury Hospital with heart failure
* NYHA functional class II-IV

Exclusion Criteria:

* Not agreeable to participate in the study
* ESRD on HD
* Severe COPD (O2/steroid dependent?)
* Pregnancy
* Hospice patients/bed bound patients
* Severe valvular disease, or recent valvular intervention (within 1 year) or planned valvular intervention.
* Expected to be transferred to another acute care hospital
* Solid organ transplant recipient or listed for transplant, recipient of left ventricular assist device or planned to receive one
* Homeless participants
* Active psychiatric disorders, addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Rate of hospital readmission for heart failure | 45 days after enrollment

SECONDARY OUTCOMES:
Quality of life: questioninaire | 45 days after enrollment
  Quality of life based on Minnesota Living with Heart Failure Questionnaire, Range 0-105, from best to worst quality of life. First time given at time of enrollment and then 45 days after enrollment, a member of the research team contacted patient by phone to complete the questionnaire.
Perceived effect of the intervention on heart-failure related care | 45 days after enrollment
  Perceived effect of the intervention on heart-failure related care based on the Perceived effect of telemonitoring questionnaire. 45 days after enrollment, a member of the research team contacted patient by phone to complete the following questions :
  1. Felt more in the control of the disease
  2. Felt more connected with the medical team
  3. Felt that it reminded to take the pills
  Each question is answered on the following scale: very true, true, somewhat true, and not true at all.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Galin, MD, Principal Investigator — Danbury Hospital, Nuvance Health
Locations (1):
- Danbury Hospital, Danbury, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No